CLINICAL TRIAL: NCT04853277
Title: Effect of Patient Education Regarding Emotional Stressors on Patient Reported Outcomes in Patients Undergoing Cellular Therapy (HSCT or CAR-T)
Brief Title: Patient Reported Outcomes and Patient Education in Cellular Therapy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Kenneth Meehan, Staff Physician, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY02000641
Record Dates: First submitted 2021-04-13; First posted 2021-04-21 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Stem Cell Transplant; CAR T-Cell Transplant; CAR T-Cell Therapy; Cellular Therapy; Hematopoietic Stem Cell Transplant; HSCT; Multiple Myeloma; Leukemia; Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Leukemia; Lymphoma | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Education Group (Experimental): Participants will receive an educational intervention focusing on psychosocial stressors and timeline of symptoms associated with the transplant/CAR-T experience.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Each Patient will undergo a 30 minute telephone visit with a trained Medical Provider outlining the timeline of various common emotional challenges experienced after transplant/CAR-T, as well as coping techniques. A pamphlet with information discussed will also be provided to the patient to review on their own time. The patient will have an opportunity to express any psychosocial/emotional concerns at this time.

SUMMARY:
The purpose of this research is to provide an educational visit addressing common emotional stressors involved in the transplant/CAR-T process, and determine if this added education improves levels of anxiety, depression, and fatigue after transplant/CART in comparison to people who do not receive the brief educational visit.

DETAILED DESCRIPTION:
Individuals who decide to participate in this study, will be provided with a survey evaluating current symptoms. This survey should take approximately 10 minutes to complete.

Individuals will then be scheduled for a 30 minute telephone visit to review common emotional stressors experienced after Stem Cell Transplant/CAR-T therapy as well as strategies to help reduce these symptoms. Participants will be provided with a pamphlet to review during the visit and independently afterwards. This visit will be conducted by telephone to avoid extra travel to the hospital, and will be conducted prior to admission for Transplant/CAR-T.

Individuals will then be asked to fill out the same set of surveys at 1 month, 3 months, 6 months, and 12 months after receiving the transplant/CAR-T therapy. These surveys will be conducted during other scheduled clinic visits to avoid additional travel to the hospital.

An individual's involvement will be complete at 1 year.

If an individual receives post-transplant/CAR-T care at a hospital other than DHMC, surveys will be mailed to the participant to complete and return at the same time points.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with an underlying hematologic disease planning to undergo an autologous or allogeneic hematopoietic stem cell transplant (HSCT) or chimeric antigen receptor T-cell (CAR-T) therapy at Dartmouth-Hitchcock Medical Center is eligible.
* The patient must be approved for HSCT/CAR-T by the treating transplant physician.

This includes completion of their pre-treatment work up and consent as directed by the standard DHMC SOPs.

- Age >18 years, and no upper age limit

Exclusion Criteria:

* Any patient with medical, social, or psychological factors that would prevent the patient from cooperating with the trial and completing surveys at requested intervals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-02-07 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Change in levels of anxiety, depression, and fatigue as measured by PROMIS-29 | Baseline (pre-transplant) and 1, 3, 6, and 12-months post-transplant/CAR-T
  Patient-Reported Outcomes Measurement Information System (PROMIS-29) includes 29 questions for 8 categories (Physical Function, Anxiety, Depression, Fatigue, Sleep Disturbance, Ability to Participate in Social Roles and Activities, Pain Interference, and Pain Intensity) with a Likert scale from 1-5. Transformed scores will be used in analysis. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. For the categories measured in this study (Anxiety, Depression, and Fatigue) a higher value represents greater symptom burden, while a lower value represents lower symptom burden.
Change in levels of anxiety, depression, and fatigue as measured by NCCN Distress Thermometer | Baseline (pre-transplant) and 1, 3, 6, and 12-months post-transplant/CAR-T
  The National Comprehensive Cancer Network (NCCN) Thermometer consists of a single-item self-report measure of psychological distress, which consists of an 11-point scale with the endpoints labeled "No distress" (0) and "Extreme distress" (10).

SECONDARY OUTCOMES:
Overall Survival | 12-months post-transplant
Post-Transplant Complications | Day 0 (date cells are infused) to 12-months post-transplant
  Post-transplant complications are defined as infections, hospitalizations, and graft versus host disease (GVHD).

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
At this time there are no plans to share IPD.